CLINICAL TRIAL: NCT06207383
Title: Catheter ABlation of Atrial Fibrillation Versus Atrioventricular Nodal Ablation with CondUction System Pacing in Persistent Atrial Fibrillation and Heart Failure
Brief Title: Atrial Fibrillation Ablation Versus Atrioventricular Nodal Ablation with Conduction System Pacing in Heart Failure
Acronym: ABACUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Haran Burri, MD, Chief Investigator and Sponsor Representative, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNF_32003B_220116
Record Dates: First submitted 2023-12-17; First posted 2024-01-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation, Persistent; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atrial fibrillation ablation (Other): Catheter ablation of atrial fibrillation using technique at the investigator's discretion but including pulmonary vein isolation as an endpoint.
  Interventions: Procedure: Atrial fibrillation ablation
- Conduction system pacing + atrioventricular nodal ablation (Active Comparator): Conduction system pacing (either His bundle pacing or left bundle branch area pacing) with catheter ablation of the atrioventricular node.
  Interventions: Device: Conduction system pacing; Procedure: Atrioventricular nodal ablation

INTERVENTIONS:
Device: Conduction system pacing — Conduction system pacing (either His bundle pacing or left bundle branch area pacing)
  Arms: Conduction system pacing + atrioventricular nodal ablation
Procedure: Atrioventricular nodal ablation — Catheter ablation of the atrioventricular node
  Arms: Conduction system pacing + atrioventricular nodal ablation
Procedure: Atrial fibrillation ablation — Catheter ablation of atrial fibrillation with pulmonary vein isolation (using technique of operator's choice, with additional lesions if deemed necessary)
  Arms: Atrial fibrillation ablation

SUMMARY:
The goal of this clinical trial is to evaluate two treatment strategies in patients with chronic atrial fibrillation and heart failure, who are eligible for atrial fibrillation ablation. Patients will be randomized to either atrial fibrillation ablation or to implantation of a pacemaker with conduction system pacing followed by atrioventricular node ablation. The effect of treatment allocation on total mortality, cardiovascular hospitalization and heart failure hospitalization will be compared.

DETAILED DESCRIPTION:
Aim To compare clinical outcome with a strategy of conduction system pacing and atrioventricular nodal ablation (CSP+AVNA), versus atrial fibrillation (AF) ablation by pulmonary vein isolation (PVI) in patients with persistent atrial fibrillation (AF) and heart failure (HF), to guide future management of these patients.

Hypotheses

1. CSP+AVNA is superior to AF ablation in patients with persistent AF and HF for reducing mortality and cardiovascular hospitalization.
2. CSP+AVNA is non-inferior to AF ablation in patients with persistent AF for reducing mortality and heart failure hospitalization.

Design Investigator-initiated, prospective randomized, controlled, open-label, multicentre study conducted in ~ 30 centres from 14 countries in Europe with expertise in CSP and AF ablation.

Sample size 220 patients

Study duration 4 years

ELIGIBILITY:
Inclusion Criteria:

(i) Persistent AF with symptomatic HF despite medical therapy, considered to be suitable for AF ablation, with at most one previous PVI procedure.

(ii) At least one prior hospital admission, or emergency room / HF clinic visit for HF in the past 2 years, with NT-pro-BNP > 1000 pg/ml or BNP > 250 pg/ml measured at any timepoint during this interval.

(iii) Previous or current rate or rhythm control drug therapy. (iv) Age > 60 years

Exclusion Criteria:

(i) NYHA Class IV and systolic blood pressure ≤80 mmHg despite optimized therapy.

(ii) Life expectancy < 2 years. (iii) Need for major surgical intervention. (iv) Myocardial infarction, stroke or PCI within the previous 3 months. (v) Previously implanted or planned implantation of CRT device or pacemaker. Implantable cardioverter defibrillator (ICD) implantation without a pacing indication is acceptable.

(vi) Participation in another controlled trial. (vii) Inability to sign and informed consent form.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Superiority endpoint | 1-4 years
  Incidence of mortality and cardiovascular hospitalization in each arm
Non-inferiority endpoint | 1-4 years
  Incidence of mortality and heart failure hospitalization in each arm

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure quality of life measure | 1 year
  The questionnaire is comprised of 21 questions around physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. The patient marks a 0-5 scale to indicate the extent to which each itemized adversity of heart failure has prevented the patient from living as they wanted to live during the past 4 weeks. The questionnaire is scored by summation of all 21 responses (the higher the score, the worse the quality of life).
Left ventricular ejection fraction | 1 year
  Measurement using echocardiography
Complications | 1-4 years
  Peri-procedural and long-term
NYHA class | 1-4 years
  New York Heart Association classification of heart failure symptoms
Cost-Effectiveness Analysis | 1-4 years
  Evaluation of clinical outcomes and associated costs between between the study arms. This evaluation will be conducted from a societal perspective, capturing both the direct medical costs and the broader societal impacts of the interventions.

CONTACTS AND LOCATIONS:
Locations (18):
- St Elisabeth sister's Hospital, Graz, Austria
- Antwerp University Hospital, Antwerp, Belgium
- Acibadem City Clinic Tokuda University Hospital, Sofia, Bulgaria
- University Hospital, Kralovske Vinohrady, Prague, Czechia
- Heart and Lung Center, University of Helsinki, Helsinki, Finland
- Hôpital Charles Nicolle, Rouen, France
- Herzzentrum Leipzig, Leipzig, Germany
- Semmelweis University, Budapest, Hungary
- Bologna University Hospital, Bologna, Italy
- University Hospital Maastricht, Maastricht, Netherlands
- Jagiellonian University, Krakow, Poland
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario y Politecnico La Fe, Madrid
- Switzerland (4):
  - University Hospital Geneva, Geneva, Canton of Geneva
  - University Hospital of Basel, Basel
  - Inselspital, Bern
  - University Hospital of Zurich, Zurich
- National Heart and Lung Institute, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data repository
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study closure
Access Criteria: Request to study P.I.